CLINICAL TRIAL: NCT07382427
Title: A Phase 2, Randomized, Single-blind, Active- and Vehicle-controlled Study to Assess the Safety, Tolerability, and Efficacy of 2.4% Terbinafine Hydrochloride Topical Solution (AP4500) in Participants With Mild to Moderate Onychomycosis of the Toenails
Brief Title: A Phase 2 Study to Assess the Effectiveness of Topical Terbinafine in Participants With Mild to Moderate Onychomycosis of the Toenails
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Onyx Axiom (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ONX-001
Record Dates: First submitted 2025-11-20; First posted 2026-02-02 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Onychomycosis of Toenail
MeSH Terms: interventions — Terbinafine; efinaconazole

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (5):
- 2.4% Topical Terbinafine once per day (Experimental): Novel topical terbinafine formulation developed to increase drug absorption through the nail. Applied once per day.
  Interventions: Drug: 2.4% Topical Terbinafine
- 2.4% Topical Terbinafine twice per day (Experimental): Novel topical terbinafine formulation developed to increase drug absorption through the nail. Applied twice per day.
  Interventions: Drug: 2.4% Topical Terbinafine
- 10% Topical Efinaconazole once per day (Active Comparator): Commercial comparator product approved for the treatment of onychomycosis. Applied once per day, as per labelled instructions.
  Interventions: Drug: 10% Topical Efinaconazole
- Topical Vehicle once per day (Placebo Comparator): Vehicle formulation without drug to act as control group for the experimental product. Applied once per day.
  Interventions: Other: Vehicle Control
- Topical Vehicle twice per day (Placebo Comparator): Vehicle formulation without drug to act as control group for the experimental product. Applied twice per day.
  Interventions: Other: Vehicle Control

INTERVENTIONS:
Drug: 2.4% Topical Terbinafine — Novel topical terbinafine product designed to increase terbinafine absorption through the nail to the site of infection
  Arms: 2.4% Topical Terbinafine once per day; 2.4% Topical Terbinafine twice per day
Drug: 10% Topical Efinaconazole — Commercial topical efinaconazole formulation approved for the treatment of onychomycosis
  Arms: 10% Topical Efinaconazole once per day
Other: Vehicle Control — Vehicle control formulation to act as a control for the experimental product
  Arms: Topical Vehicle once per day; Topical Vehicle twice per day

SUMMARY:
Onychomycosis is a fungal infection of the toenail caused by a range of organisms, including dermophytes, non-dermophyte molds, and yeasts. Topical antifungals are often used for mild to moderate onychomycosis, especially when oral therapy is contraindicated. Generally, topical antifungal agents are well-tolerated with minimal side effects, but they are less effective than oral antifungal therapies due to poor nail penetration. Consequently, the current treatment period for topical onychomycosis products is ~12 months.

Terbinafine is an antifungal drug approved by the FDA for the treatment of topical skin infections. A new formulation (AP4500) has been developed to increase terbinafine absorption through the nail in order to directly kill fungi at the site of onychomycosis infection.

The goal of this clinical trial is to learn if AP4500 works to treat mild to moderate toenail fungus in adults. The main questions the study aims to answer are:

Does AP4500 work to treat onychomycosis? Does AP4500 work best when applied once or twice per day? Does AP4500 treat onychomycosis faster than current treatments? Is AP4500 more effective than current treatments?

Researchers will compare AP4500 to a vehicle control (a look-alike substance that contains no drug) and a commercial comparator product (Jublia) that has already been commercialized for the treatment of toenail fungus.

Participants will:

Apply topical formulations once or twice a day to an infected toenail for a period of 48 weeks Visit the clinic 4 times over this period for checkups and tests, with a subsequent follow up visit 4 weeks after treatment is completed

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants aged 18 to 70 years, inclusive at the time of informed consent.
* In general, good health, as assessed by the Investigator, as determined by medical history, safety laboratory tests, and other tests.
* At least 1 great toenail (the "target great toenail") with clinically diagnosed distal lateral subungual onychomycosis involving 20% to 50% of the affected great toenail but with no more than 6 toenails and no fingernails involved, and without dermatophytomas or lanula (matrix) involvement.
* Target great toenail must have an uninfected length of at least 3 mm from the proximal nailfold and a thickness of no more than 3 mm.
* Target great toenail must have evidence of toenail growth per the participant's report that monthly clipping is required.
* Within 42 days prior to Baseline (Day 1), must have a positive potassium hydroxide (KOH) examination of the target great toenail.
* Within 42 days prior to Baseline (Day 1), must have a positive dermatophyte culture for Trichophyton rubrum or Trichophyton mentagrophytes from the target great toenail.
* Women of childbearing potential (WOCBP) must have a negative pregnancy test at Screening and prior to dosing and be willing to have additional pregnancy tests as required throughout the trial. Women not of childbearing potential are women who are either permanent sterile or postmenopausal. Permanent sterilization methods include hysterectomy, bilateral salpingectomy and bilateral oophorectomy. A postmenopausal state is defined as no menses for 12 months without an alternative medical cause. Postmenopausal status will be confirmed through testing of follicle-stimulating hormone (FSH) levels ≥40 IU/L at Screening for amenorrheic female participants.
* Agree to avoid the use of toenail polish, cosmetic toenail products, and pedicures during the trial period.
* Written informed consent from the participant prior to any trial procedures.
* Willing and able to comply with the scheduled visits, confinement period, treatment plan, laboratory tests, and other trial procedures and requirements.

Exclusion Criteria:

* Presence of any toenail infection other than or in addition to dermatophytes, such as Scytalidium as determined by the Investigator (candidal onychomycosis infection, concurrent with a positive dermatophyte culture, is acceptable).
* Presence of any of the following: dermatophytoma, fungal "spikes" within 3 mm of the proximal toenail fold on the target great toenail, infection extending to the matrix, or only lateral toenail disease in the target great toenail.
* Presence of severe moccasin tinea pedis at the Screening or Baseline visits, as determined by the Investigator. If the participant has interdigital tinea pedis that requires treatment, the participant must agree to use only an Investigator-approved topical antifungal therapy .
* Presence of any disease/condition that might cause toenail abnormalities or may interfere with the evaluation of the investigational medicinal product (IMP), as determined by the Investigator (e.g., open sore or ulceration on the toes of affected toenails, psoriasis, immune dysfunction immunocompromised, collagen-vascular diseases, lichen planus, peripheral vascular disease, recurrent cellulitis, lymphatic insufficiency, or traumatic onychodystrophy due to chronic physical stimuli).
* Any previous surgery on the target great toenail.
* Presence of onychomycosis of the fingernail or fingernail dermatophytosis.
* Target great toenail (including the toenail plate and any subungual debris) thicker than 3 mm at the Screening and Baseline visit - Day 1s.
* Presence of onychodystrophy that could interfere with clinical assessments, as determined by the Investigator.
* Presence of any underlying disease or dermatological condition that, in the opinion of the Investigator, could present a safety concern for the participant or that could interfere with clinical evaluations.
* Use of the following topical preparations within the indicated time prior to the Baseline visit (Day 1) or need for concurrent use of any of the following topical preparations during the trial; Toenail polish or cosmetic toenail products: 1 day; Other topical prescription or over-the-counter medications to the toenails (with the exception of bland emollients): 2 weeks; Topical prescription or over-the-counter antifungal therapy for the toenails, including devices to treat onychomycosis: 4 weeks
* Use of the following systemic medications within the indicated time prior to the Baseline visit or need for concurrent use of any of the following systemic medications during the trial; Systemic antifungal therapy: 4 weeks; Systemic immunosuppressive agents: 6 months; History of oral antifungal with known activity against dermatophytes within twelve months prior to Screening.
* Known human immunodeficiency virus (HIV) infection self-reported or as determined by the Investigator.
* Received treatment for any type of cancer in the previous 6 months, with the exception of nonmelanoma skin cancer (e.g., basal cell carcinoma or nonmetastatic squamous cell carcinoma) that was treated successfully .
* Diagnosis of diabetes mellitus.
* History of hypersensitivity or allergic reactions to any of the IMP constituents.
* Females who are pregnant, lactating, or planning a pregnancy during the trial period.
* History of immunosuppression and/or clinical signs indicative of possible immunosuppression, as determined by the Investigator.
* History of drug abuse or addiction in the last 12 months of enrolment that, in the opinion of the Investigator, could affect the participant's safety and/or compliance with the trial .
* History of alcohol abuse that, in the opinion of the Investigator, could affect the participant's safety and/or compliance with the trial. As per Australian Alcohol Guidelines, Australian Government it is recommended regular consumption of more than 10 standard drinks/week and/or no more than 4 standard drinks on any single day, where 1 standard drink is 10 g of pure alcohol and is equivalent to 285mL beer (4.9% alcohol/volume), 100 mL wine (12% alcohol/volume) or 30 mL spirit (40% alcohol/volume).

Use of any investigational drug or device within 30 days of 5 half-lives (whichever is longer) prior to the Screening visit or concurrent participation in another clinical trial with an investigational drug or device.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2028-01 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Number of patients with Complete Cure at Weeks 12, 24, 36, 48, and 52 | 52 weeks
  Complete Cure is defined as 0% visible onychomycosis of the target great toenail upon examination and negative potassium hydroxide [KOH] fungal culture

SECONDARY OUTCOMES:
Number of participants with Almost Complete Cure at Weeks 12, 24, 36, 48 and 52 | 52 weeks
  Almost Complete Cure defined as onychomycosis affecting a maximum of 5% toenail after visual examination and negative KOH examination and fungal culture
Incidence, severity, and relationship to treatment of treatment emergent adverse events (TEAEs), serious adverse events (SAEs), and adverse events (AEs) as coded by MedDRA | 52 weeks
  A by participate adverse event data listing, including verbatim term, preferred term, system organ class, severity, and relationship to the investigational medicinal product are to be provided.
Time to Clinical Efficacy in participants over 48 weeks | 52 weeks
  Affected toenails will be visually assessed at 12, 24, 36, 48 and 52 weeks for Clinical Efficacy (defined as a maximum of 10% of the nail demonstrating onychomycosis)

IPD SHARING:
Plan to Share IPD: No
This is an industry sponsored trial using a proprietary formulation. Results will be commercially confidential.